CLINICAL TRIAL: NCT02815397
Title: DA-EPOCH-RM: A Phase II Study Evaluating the Efficacy and Safety of Metformin in Combination With Standard Induction Therapy (DA-EPOCH-R) for Previously Untreated C-myc+ Diffuse Large B-Cell Lymphoma
Brief Title: DA-EPOCH-Rituximab/Metformin (RM) for Double Hit Lymphoma
Acronym: DLBCL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Rush University Medical Center (Other)
Collaborators: Elsa U. Pardee Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYM15 DA-EPOCH-RM
Record Dates: First submitted 2016-05-17; First posted 2016-06-28 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2016-12

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Double Hit DLBCL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm, open label (Experimental): Metformin added to standard of care treatment for all patients
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — given in addition to standard of care treatment
  Other Names: Glumetza, Fortamet, Glucophage, Riomet

SUMMARY:
Newly diagnosed histologically confirmed c-myc+ de novo DLBCL. Metformin 500 mg daily x 1 week, then 500 mg twice daily (BID) x 2 weeks, then 850 mg twice daily until 1 month after last cycle of chemo-immunotherapy.

DA-EPOCH-R every 21 days x 4 cycles (CNS prophylaxis single or triple therapy given intrathecally each cycle to patients deemed appropriate by treating physician).

Restage after 4 cycles with CT. Complete remission or partial remission: complete 2 more cycles or radiation therapy (XRT) consolidation per physician. Stable or progressive disease will go on to salvage therapy off study.

DETAILED DESCRIPTION:
Subject admitted to in-patient care for day 1 or each cycle and discharged on day 5. On day 6, subject receives Rituximab in outpatient infusion facility.

Metformin is dispensed on day 1 of each cycle and taken as follows: Cycle 1 days 1-7 500 mg daily. Days 8-21, 500 mg twice daily. Cycle 2 through end of treatment, metformin given 850 mg twice daily.

Inpatient treatment: DA-EPOCH every 21 days Etoposide (VP-16) 50 mg/m2/d civi d1-4 (continuous infusion) Prednisone 60 mg/m2 BID po d1-5 Vincristine 0.4 mg/m2/d civi d 1-4 (continuous infusion) Doxorubicin (Adriamycin) 10 mg/m2/d civi d1-4 (continuous infusion) Cyclophosphamide (Cytoxan) 750 mg/m2 IV over 15 min d5 If clinically indicated, patients who are deemed appropriate for central nervous system (CNS) prophylaxis by their treating physician will receive either single agent intrathecal methotrexate (12 mg) or triple therapy (15 mg methotrexate, 30 mg cytarabine, 30 mg hydrocortisone) with each cycle of chemotherapy.

Rituximab 375 mg/m2 IV every 21 days on D6-8 post DA-EPOCH (per standard institutional guidelines) DA-dose adjustment paradigm based on twice weekly complete blood count (CBC) (dose adjustment above starting doses apply to Etoposide (VP-16), Doxorubicin (Adriamycin) and Cyclophosphamide (Cytoxan). If nadir absolute neutrophil count(ANC)>500/microliter (uL), 20% increase in all 3 drugs. If nadir<500/uL on 1 or 2 measurements, same doses as last cycle. If nadir <500/uL on at least 3 measurements, or nadir platelet <25,000/uL on 1 measurement, 20% decrease in Etoposide, Doxorubicin and Cyclophosphamide below last cycle.

Filgrastim (Neupogen) 5 mcg/kg sc qd beginning on d6 until ANC>5,000/uL or Pegfilgrastim (Neulasta) 6 mg sc 24-72 hours post chemotherapy.

Restaging with CT scans is done after cycle 4 and:

complete remission (CR)/partial remission (PR) - complete 2 more cycles of therapy OR consolidation radiation therapy per treating physician.

stable disease (SD)/progressive disease (PD) - salvage therapy off study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Diagnosis of DLBCL as documented by medical records and with histology based on criteria established by the World Health Organization

  * subtyping is required for DLBCL
  * c-myc+ defined as presence of c-myc breaks by karyotype/FISH and/or IHC ≥ 40%; this includes double hits (with bcl-2 breaks found using cytogenetics/FISH) and/or double expressors (with bcl-2 protein expression ≥ 70% by IHC); increased copy number in itself is not considered positivity for c-myc
* No prior therapy for diagnosis of DLBCL with exception of steroids
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0- 2 (Appendix B)
* Life expectancy of at least 6 months
* No history of medication dependent diabetes mellitus
* No evidence of acute or chronic metabolic acidosis (baseline venous lactate ≤ 4)

Exclusion Criteria

* Patient already on any class of anti-diabetic medication including metformin, insulin analogues, sulfonylureas, thiazolidinediones (TZDs) and the incretin-based therapies or clear need for therapeutic intervention based on fasting blood glucose
* Known histological transformation from indolent non-Hodgkin Lymphoma (iNHL) or chronic lymphocytic leukemia (CLL) to an aggressive form of non-Hodgkin's lymphoma (NHL) (ie, Richter transformation)
* Burkitt and/or precursor lymphoblastic leukemia/lymphoma.
* Presence of known intermediate- or high-grade myelodysplastic syndrome
* History of an active of treated non-lymphoid malignancy within the last 3 years excluding basal cell and squamous cell skin cancers
* Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of start of study drug.
* Subjects who have currently active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver involvement with NHL or stable chronic liver disease per investigator assessment)
* Renal insufficiency with creatinine > 1.5 x upper limit of normal (ULN) OR creatinine clearance of < 45 ml/min as calculated by the Cockcroft-Gault method
* CNS or leptomeningeal involvement of lymphoma
* HIV positive
* Ongoing inflammatory bowel disease
* Ongoing alcohol or drug addiction
* Pregnancy or breastfeeding
* History of prior allogeneic bone marrow progenitor cell or solid organ transplantation -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reem Karmali, MD, Principal Investigator — Rush Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm, Open Label
Started | 2
Completed | 0
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm, Open Label
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Impact of Metformin on 18 Month Progression-free Survival
Description: Progression-free survival determined by CT scans at 18 months
Time Frame: 18 month
Population: will not have this data as study closed prematurely.
Arm/Group | Single Arm, Open Label
Number analyzed (Participants) | 0

2. Secondary Outcome: Effect of Metformin Overall Response Rate
Description: Evaluation of the effect of the addition of metformin to induction chemotherapy on overall response rates
Time Frame: 3 years
Population: no data available as study closed before response could be determined
Arm/Group | Single Arm, Open Label
Number analyzed (Participants) | 0

3. Secondary Outcome: Effect of Metformin Overall Survival
Description: Evaluation of the addition of metformin to standard induction therapy on 18 month overall survival
Time Frame: 18 months
Population: will not have this data as study closed prematurely.
Arm/Group | Single Arm, Open Label
Number analyzed (Participants) | 0

4. Secondary Outcome: Safety Profile With Addition of Metformin Evaluated by Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v.4.0
Description: Describe the safety profile observed by measuring fasting glucose and anion gap weekly through cycle 6.
Time Frame: 18 months
Population: will not have this data as study closed prematurely.
Arm/Group | Single Arm, Open Label
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Trial closed prematurely - adverse event data not collected
Description: Serious and Other [Not Including Serious] Adverse Events were not collected/assessed
Arm/Group | Single Arm, Open Label
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Study closed prematurely - will not be able to report on any PFS, OS, ORR. Will not have any additional information on adverse events/toxicity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes